CLINICAL TRIAL: NCT03200639
Title: Comparison of High Intensity Interval Body Weight Training Versus Combined Training on Body Composition, Physical Function, Metabolic Risk and Inflammation in Postmenopausal Women With and Without Gynecological Cancer
Brief Title: Cachexia in Gynecological Cancer and the Preventive Role of Weight Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Triangulo Mineiro (Other)
Responsible Party: Principal Investigator, Fábio Lera Orsatti, Professor, PhD, Universidade Federal do Triangulo Mineiro
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CAAE: 45108115.8.0000.5154
Record Dates: First submitted 2017-06-20; First posted 2017-06-27 (Actual); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Breast Cancer Female; Gynecologic Cancer; Menopause; Physical Activity
Keywords: Breast Cancer Female; Gynecologic Cancer; Menopause; Physical Activity
MeSH Terms: conditions — Motor Activity | interventions — High-Intensity Interval Training; Weights and Measures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Physical training, CT (Active Comparator): Combined Trained with no cancer (CT): Post menopausal women with no cancer submitted to 12 weeks of combined training (i.e. aerobic training plus resistance training)
  Interventions: Other: Combined training
- Physical training, HIITBW (Active Comparator): High intensity interval training with body weight with no cancer (HIITBW): Post menopausal women with no cancer submitted to 12 weeks of high intensity interval training with body weight (i.e. step climbing plus squats)
  Interventions: Other: High intensity interval training with body weight
- Physical training, CTc (Experimental): Combined Trained with gynecological and/or breast cancer (CTc): Post menopausal women with with gynecological and/or breast cancer submitted to 12 weeks of combined training (i.e. aerobic training plus resistance training)
  Interventions: Other: Combined training
- Physical training, HIITBWc (Experimental): High intensity interval training with body weight with gynecological and/or breast cancer (HIITBWc): Post menopausal women with gynecological and/or breast cancer submitted to 12 weeks of high intensity interval training with body weight (i.e. step climbing plus squats)
  Interventions: Other: High intensity interval training with body weight

INTERVENTIONS:
Other: Combined training — The CT and CTc protocol (total length time ~60 min) were performed three times a week for 12 weeks, in nonconsecutive days, and were composed by 30-min walk at 70% of maximum heart rate or Borg Scale at 5-6 following resistance exercises (RE: 45-degree half squat, bench press, leg curl, rowing machine and unilateral leg extension) at 70% of one repetition maximum (1RM) with three sets of 8-12 repetitions and 1.5 min rest interval between sets and exercises. If the volunteer exceeded or did not reach the walk intensity, the volunteer was stimulated by to decrease or increase the walk speed, respectively. Regarding the resistance exercises, the load was adjusted in the 6th week with the 1RM test to ensure the 70% of 1RM between 8-12 repetitions.
  Arms: Physical training, CT; Physical training, CTc
Other: High intensity interval training with body weight — The HIITBW and HIITBWc protocol (total length time ~28 min) were performed three times a week for 12 weeks, in nonconsecutive days, and were composed by ten sets of 60 s of high (vigorous) intensity exercises at 80-95% of HRmax or Borg Scale at 8-9 (i.e. 30s of stepping up and down on a step and 30s of squatting up and down as fast as possible) interspersed with a recovery of 60 s of light walk (<60% of HRmax or Borg Scale at <5). To ensure vigorous zone of all sets, if the volunteer exceeded or did not reach the vigorous zone the volunteer was stimulated by the fitness professionals to decrease or increase the number of steps and squats, respectively.
  Arms: Physical training, HIITBW; Physical training, HIITBWc

SUMMARY:
The study aim was to compare the effectiveness of combined training (CT; aerobic + resistance exercises) and high-intensity interval body weight training (HIITBW) on body composition, metabolic and inflammatory profile, physical function and quality of life in older women with gynecological and breast cancer and their pair-matched controls (older women with no cancer). The hypothesis of the present clinical trial is that HIITBW is effective as well as CT for improvements on body composition, metabolic and inflammatory profile, physical function and quality of life in older women with gynecological and breast cancer.

DETAILED DESCRIPTION:
Physical training has been recommended to prevent or attenuation cachexia and sarcopenia in older people with or without cancer. The American College of Sports Medicine recommends 150 min of moderate intensity exercise combining aerobic exercise with resistance exercises, termed as combined training (CT). However, it has been reported that very low proportion (<10%) of older adults meet the physical activity recommendation. Lack of time has been reported as a common reason to people not to do exercise. Thus, identifying effective physical training dosages and modalities which may be feasible are necessary for this population.

Repeated brief bouts of fast and intense exercise interspersed with low intensity exercise termed as high intensity interval training (HIIT) has shown to be a time-effective strategy to improve cardiorespiratory fitness in young and older. Moreover, HIIT has shown to improve glycemic control in patients at high risk for TDM2, muscle mass, body fat and physical function. However, there were many pending issues involving the HIIT for sarcopenia and cachexia in older people. For instance, the lack of access to physical activity facilities, such as the need for specific equipment (i.e. fitness equipment: treadmill, bike or resistance exercise equipment) and the need for high motor skill levels to performance the high-intensity exercise (i.e. run at high speed) have been reported as another reason to older people not to do HIIT.

Different HIIT programs performed outside of laboratory has been proposed, especially with body-weight exercises. The high-intensity interval body weight training (HIBWT) is performed without equipment and with low motor skill levels. HIBWT has been shown to improve fat mass, muscle mass, cardiorespiratory capacity and physical performance in young adults with or without overweight. Despite this, no previous studies have evaluated HIBWT efficacy and safe in older people with sarcopenia and cachexia. The study aim was to compare the effectiveness of CT and HIITBW on body composition, metabolic and inflammatory profile, physical function and quality of life in older women with gynecological and breast cancer and their pair-matched controls (older women with no cancer). The hypothesis of the present clinical trial is that HIITBW is effective as well as CT for improvements on body composition, metabolic and inflammatory profile, physical function and quality of life in older women with gynecological and breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Postemenopausal women without cancer
* Postemenopausal women with breast cancer
* Postemenopausal women with gynecological cancer

Exclusion Criteria:

• No several physical limitations (wheelchair, canes or any similar device)

Min Age: 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2015-05-30 (Actual); Primary Completion 2015-12-01 (Actual); Study Completion 2015-12-10 (Actual)

PRIMARY OUTCOMES:
Body composition | pre intervention and post intervention (i.e. 12 weeks)
  Soft-tissue (fat mass, kg and lean mass, kg) of whole body and regional composition were assessed via dual-energy x-ray absorptiometry scanning (iDXA; GE Healthcare-Luna, Madison, WI; software Encore version 14.10)
Muscle strength | pre intervention and post intervention (i.e. 12 weeks)
  It was measured by the one repetition maximum (1RM) test in the leg extension equipment.
Rate of force development (a critical component of muscle power) | pre intervention and post intervention (i.e. 12 weeks)
  It was measured by a rapid maximum isometric voluntary contraction of the one-sidedly knee extension force pulses (Metrolog SD20-LVDT, São Carlos/SP, Brazil) of both legs.
Cardiorespiratory fitness | pre intervention and post intervention (i.e. 12 weeks)
  The six-minute walk test and the one mile walk test was performed indoor, on a flat floor in a sports court.
Short physical performance battery (SPPB) | pre intervention and post intervention (i.e. 12 weeks)
  The SPPB consisted of three tests performed in the following order: balance test, four-meter walk test, and five-time-sit-to-stand test.
  Each test score varied to zero to four points, and the SPPB total score varied to zero to 12 points (sum of the scores of the three tests).

SECONDARY OUTCOMES:
Citokines | pre intervention and post intervention (i.e. 12 weeks)
  Blood samples (16 ml) were collected between 7:30 AM and 9:00 AM after an overnight fast (10-12 hours). The blood samples (venous) were collected by a dry tube with gel separator or EDTA (vacuum-sealed system; Vacutainer, England). The sample was centrifuged for 10 minutes (3.000 rpm) and samples were separated and stocked (-80 C) for futures analysis.
  The blood indicators were measured as follows: IL-10, IL-6, IL-1ra, TNF-α, ICAM-1, MCP-1, Leptin and Total Adiponectin (enzyme-linked immunosorbent assay method) with Readwell Touch equipment (Robonik, India) and R&D kits (USA).
Quality of life | pre intervention and post intervention (i.e. 12 weeks)
  Quality of life - The 36-Item Short Form Health Survey (SF-36) was used to measure the overall quality of life aspects, separated in the following domains: functional capacity, physical limitations, pain, overall health, vitality, social aspects, emotional limitations and mental health.
Hormones | pre intervention and post intervention (i.e. 12 weeks)
  Blood samples (16 ml) were collected between 7:30 AM and 9:00 AM after an overnight fast (10-12 hours). The blood samples (venous) were collected by a dry tube with gel separator or EDTA (vacuum-sealed system; Vacutainer, England). The sample was centrifuged for 10 minutes (3.000 rpm) and samples were separated and stocked (-80 C) for futures analysis.
  The blood indicators were measured as follows: Testosterone, LH, TSH, T4, insulin, DHEA-S, E2 and FSH (electrochemoluminescence method).
Metabolic markers | pre intervention and post intervention (i.e. 12 weeks)
  Blood samples (16 ml) were collected between 7:30 AM and 9:00 AM after an overnight fast (10-12 hours). The blood samples (venous) were collected by a dry tube with gel separator or EDTA (vacuum-sealed system; Vacutainer, England). The sample was centrifuged for 10 minutes (3.000 rpm) and samples were separated and stocked (-80 C) for futures analysis.
  The blood indicators were measured as follows: Glucose, C-reactive protein, Hb1Ac (automated colorimetric method), total cholesterol, ALT and AST (kinetic method) with Cobas 6000 equipment and Roche kit (USA).
Electromyography | pre intervention and post intervention (i.e. 12 weeks)
  Quadriceps electromyography
Physical activity level | pre intervention and post intervention (i.e. 12 weeks)
  The International Physical Activity Questionnaire (IPAQ) was used to measure the level (time spent) of physical activities of light, moderate and high intensities during the day. Also, the sitting time (minutes) per day was measured.
Nutrition habits | pre intervention and post intervention (i.e. 12 weeks)
  A three-day food record (two days in the middle of week and one on the weekend) was used to determine the energy and macronutrients (carbohydrates, proteins and fats).
Functional capacity | pre intervention and post intervention (i.e. 12 weeks)
  The activities of daily living was assessed by Lawnton and Katz scale.

CONTACTS AND LOCATIONS:
Overall Officials: Fábio Orsatti, PhD, Principal Investigator — Federal University of Triângulo Mineiro

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] American College of Sports Medicine. American College of Sports Medicine position stand. Progression models in resistance training for healthy adults. Med Sci Sports Exerc. 2009 Mar;41(3):687-708. doi: 10.1249/MSS.0b013e3181915670. PMID 19204579
- [Background] Al-Majid S, Waters H. The biological mechanisms of cancer-related skeletal muscle wasting: the role of progressive resistance exercise. Biol Res Nurs. 2008 Jul;10(1):7-20. doi: 10.1177/1099800408317345. PMID 18705151
- [Background] Bickel CS, Slade J, Mahoney E, Haddad F, Dudley GA, Adams GR. Time course of molecular responses of human skeletal muscle to acute bouts of resistance exercise. J Appl Physiol (1985). 2005 Feb;98(2):482-8. doi: 10.1152/japplphysiol.00895.2004. Epub 2004 Oct 1. PMID 15465884
- [Background] Belcastro AN, Shewchuk LD, Raj DA. Exercise-induced muscle injury: a calpain hypothesis. Mol Cell Biochem. 1998 Feb;179(1-2):135-45. doi: 10.1023/a:1006816123601. PMID 9543356
- [Background] Campos GE, Luecke TJ, Wendeln HK, Toma K, Hagerman FC, Murray TF, Ragg KE, Ratamess NA, Kraemer WJ, Staron RS. Muscular adaptations in response to three different resistance-training regimens: specificity of repetition maximum training zones. Eur J Appl Physiol. 2002 Nov;88(1-2):50-60. doi: 10.1007/s00421-002-0681-6. Epub 2002 Aug 15. PMID 12436270
- [Background] Carson JA, Baltgalvis KA. Interleukin 6 as a key regulator of muscle mass during cachexia. Exerc Sport Sci Rev. 2010 Oct;38(4):168-76. doi: 10.1097/JES.0b013e3181f44f11. PMID 20871233
- [Background] Charge SB, Rudnicki MA. Cellular and molecular regulation of muscle regeneration. Physiol Rev. 2004 Jan;84(1):209-38. doi: 10.1152/physrev.00019.2003. PMID 14715915
- [Background] Ciechanover A. The ubiquitin-proteasome pathway: on protein death and cell life. EMBO J. 1998 Dec 15;17(24):7151-60. doi: 10.1093/emboj/17.24.7151. No abstract available. PMID 9857172
- [Background] Cruz-Jentoft AJ, Baeyens JP, Bauer JM, Boirie Y, Cederholm T, Landi F, Martin FC, Michel JP, Rolland Y, Schneider SM, Topinkova E, Vandewoude M, Zamboni M; European Working Group on Sarcopenia in Older People. Sarcopenia: European consensus on definition and diagnosis: Report of the European Working Group on Sarcopenia in Older People. Age Ageing. 2010 Jul;39(4):412-23. doi: 10.1093/ageing/afq034. Epub 2010 Apr 13. PMID 20392703
- [Background] Donohoe CL, Ryan AM, Reynolds JV. Cancer cachexia: mechanisms and clinical implications. Gastroenterol Res Pract. 2011;2011:601434. doi: 10.1155/2011/601434. Epub 2011 Jun 13. PMID 21760776
- [Background] Eliakim A, Nemet D. Exercise training, physical fitness and the growth hormone-insulin-like growth factor-1 axis and cytokine balance. Med Sport Sci. 2010;55:128-140. doi: 10.1159/000321977. Epub 2010 Oct 14. PMID 20956865
- [Background] Farkas J, von Haehling S, Kalantar-Zadeh K, Morley JE, Anker SD, Lainscak M. Cachexia as a major public health problem: frequent, costly, and deadly. J Cachexia Sarcopenia Muscle. 2013 Sep;4(3):173-8. doi: 10.1007/s13539-013-0105-y. Epub 2013 Mar 29. PMID 23539127
- [Background] Fluck M, Hoppeler H. Molecular basis of skeletal muscle plasticity--from gene to form and function. Rev Physiol Biochem Pharmacol. 2003;146:159-216. doi: 10.1007/s10254-002-0004-7. Epub 2003 Jan 14. PMID 12605307
- [Background] Frystyk J. Exercise and the growth hormone-insulin-like growth factor axis. Med Sci Sports Exerc. 2010 Jan;42(1):58-66. doi: 10.1249/MSS.0b013e3181b07d2d. PMID 20010129
- [Background] Glass D, Roubenoff R. Recent advances in the biology and therapy of muscle wasting. Ann N Y Acad Sci. 2010 Nov;1211:25-36. doi: 10.1111/j.1749-6632.2010.05809.x. PMID 21062293
- [Background] Gould DW, Lahart I, Carmichael AR, Koutedakis Y, Metsios GS. Cancer cachexia prevention via physical exercise: molecular mechanisms. J Cachexia Sarcopenia Muscle. 2013 Jun;4(2):111-24. doi: 10.1007/s13539-012-0096-0. Epub 2012 Dec 13. PMID 23239116
- [Background] Hansen J, Brandt C, Nielsen AR, Hojman P, Whitham M, Febbraio MA, Pedersen BK, Plomgaard P. Exercise induces a marked increase in plasma follistatin: evidence that follistatin is a contraction-induced hepatokine. Endocrinology. 2011 Jan;152(1):164-71. doi: 10.1210/en.2010-0868. Epub 2010 Nov 10. PMID 21068158
- [Background] Hasselgren PO, Fischer JE. Muscle cachexia: current concepts of intracellular mechanisms and molecular regulation. Ann Surg. 2001 Jan;233(1):9-17. doi: 10.1097/00000658-200101000-00003. PMID 11141219
- [Background] Hawke TJ, Garry DJ. Myogenic satellite cells: physiology to molecular biology. J Appl Physiol (1985). 2001 Aug;91(2):534-51. doi: 10.1152/jappl.2001.91.2.534. PMID 11457764
- [Background] Jagoe RT, Redfern CP, Roberts RG, Gibson GJ, Goodship TH. Skeletal muscle mRNA levels for cathepsin B, but not components of the ubiquitin-proteasome pathway, are increased in patients with lung cancer referred for thoracotomy. Clin Sci (Lond). 2002 Mar;102(3):353-61. PMID 11869177
- [Background] Janssen I, Baumgartner RN, Ross R, Rosenberg IH, Roubenoff R. Skeletal muscle cutpoints associated with elevated physical disability risk in older men and women. Am J Epidemiol. 2004 Feb 15;159(4):413-21. doi: 10.1093/aje/kwh058. PMID 14769646
- [Background] Khal J, Wyke SM, Russell ST, Hine AV, Tisdale MJ. Expression of the ubiquitin-proteasome pathway and muscle loss in experimental cancer cachexia. Br J Cancer. 2005 Oct 3;93(7):774-80. doi: 10.1038/sj.bjc.6602780. PMID 16160695
- [Background] Laviano A, Meguid MM, Inui A, Muscaritoli M, Rossi-Fanelli F. Therapy insight: Cancer anorexia-cachexia syndrome--when all you can eat is yourself. Nat Clin Pract Oncol. 2005 Mar;2(3):158-65. doi: 10.1038/ncponc0112. PMID 16264909
- [Background] Lecker SH, Solomon V, Mitch WE, Goldberg AL. Muscle protein breakdown and the critical role of the ubiquitin-proteasome pathway in normal and disease states. J Nutr. 1999 Jan;129(1S Suppl):227S-237S. doi: 10.1093/jn/129.1.227S. No abstract available. PMID 9915905
- [Background] Long CL, Birkhahn RH, Geiger JW, Betts JE, Schiller WR, Blakemore WS. Urinary excretion of 3-methylhistidine: an assessment of muscle protein catabolism in adult normal subjects and during malnutrition, sepsis, and skeletal trauma. Metabolism. 1981 Aug;30(8):765-76. doi: 10.1016/0026-0495(81)90022-6. PMID 6790901
- [Background] Lowell BB, Ruderman NB, Goodman MN. Evidence that lysosomes are not involved in the degradation of myofibrillar proteins in rat skeletal muscle. Biochem J. 1986 Feb 15;234(1):237-40. doi: 10.1042/bj2340237. PMID 3707546
- [Background] Matthys P, Mitera T, Heremans H, Van Damme J, Billiau A. Anti-gamma interferon and anti-interleukin-6 antibodies affect staphylococcal enterotoxin B-induced weight loss, hypoglycemia, and cytokine release in D-galactosamine-sensitized and unsensitized mice. Infect Immun. 1995 Apr;63(4):1158-64. doi: 10.1128/iai.63.4.1158-1164.1995. PMID 7890366
- [Background] Mizuhara H, O'Neill E, Seki N, Ogawa T, Kusunoki C, Otsuka K, Satoh S, Niwa M, Senoh H, Fujiwara H. T cell activation-associated hepatic injury: mediation by tumor necrosis factors and protection by interleukin 6. J Exp Med. 1994 May 1;179(5):1529-37. doi: 10.1084/jem.179.5.1529. PMID 8163936
- [Background] Muscaritoli M, Anker SD, Argiles J, Aversa Z, Bauer JM, Biolo G, Boirie Y, Bosaeus I, Cederholm T, Costelli P, Fearon KC, Laviano A, Maggio M, Rossi Fanelli F, Schneider SM, Schols A, Sieber CC. Consensus definition of sarcopenia, cachexia and pre-cachexia: joint document elaborated by Special Interest Groups (SIG) "cachexia-anorexia in chronic wasting diseases" and "nutrition in geriatrics". Clin Nutr. 2010 Apr;29(2):154-9. doi: 10.1016/j.clnu.2009.12.004. Epub 2010 Jan 8. PMID 20060626
- [Background] Pedersen BK. Muscle as a secretory organ. Compr Physiol. 2013 Jul;3(3):1337-62. doi: 10.1002/cphy.c120033. PMID 23897689
- [Background] Pedersen BK, Febbraio MA. Muscles, exercise and obesity: skeletal muscle as a secretory organ. Nat Rev Endocrinol. 2012 Apr 3;8(8):457-65. doi: 10.1038/nrendo.2012.49. PMID 22473333
- [Background] Pette D, Staron RS. Transitions of muscle fiber phenotypic profiles. Histochem Cell Biol. 2001 May;115(5):359-72. doi: 10.1007/s004180100268. PMID 11449884
- [Background] Pickering WP, Price SR, Bircher G, Marinovic AC, Mitch WE, Walls J. Nutrition in CAPD: serum bicarbonate and the ubiquitin-proteasome system in muscle. Kidney Int. 2002 Apr;61(4):1286-92. doi: 10.1046/j.1523-1755.2002.00276.x. PMID 11918735
- [Background] Rall LC, Roubenoff R. Rheumatoid cachexia: metabolic abnormalities, mechanisms and interventions. Rheumatology (Oxford). 2004 Oct;43(10):1219-23. doi: 10.1093/rheumatology/keh321. Epub 2004 Aug 3. PMID 15292530
- [Background] Schakman O, Gilson H, Kalista S, Thissen JP. Mechanisms of muscle atrophy induced by glucocorticoids. Horm Res. 2009 Nov;72 Suppl 1:36-41. doi: 10.1159/000229762. Epub 2009 Nov 27. PMID 19940494
- [Background] Schakman O, Kalista S, Barbe C, Loumaye A, Thissen JP. Glucocorticoid-induced skeletal muscle atrophy. Int J Biochem Cell Biol. 2013 Oct;45(10):2163-72. doi: 10.1016/j.biocel.2013.05.036. Epub 2013 Jun 24. PMID 23806868
- [Background] Seale P, Rudnicki MA. A new look at the origin, function, and "stem-cell" status of muscle satellite cells. Dev Biol. 2000 Feb 15;218(2):115-24. doi: 10.1006/dbio.1999.9565. PMID 10656756
- [Background] Serrano AL, Baeza-Raja B, Perdiguero E, Jardi M, Munoz-Canoves P. Interleukin-6 is an essential regulator of satellite cell-mediated skeletal muscle hypertrophy. Cell Metab. 2008 Jan;7(1):33-44. doi: 10.1016/j.cmet.2007.11.011. PMID 18177723
- [Background] Spiering BA, Kraemer WJ, Anderson JM, Armstrong LE, Nindl BC, Volek JS, Maresh CM. Resistance exercise biology: manipulation of resistance exercise programme variables determines the responses of cellular and molecular signalling pathways. Sports Med. 2008;38(7):527-40. doi: 10.2165/00007256-200838070-00001. PMID 18557656
- [Background] Starkie R, Ostrowski SR, Jauffred S, Febbraio M, Pedersen BK. Exercise and IL-6 infusion inhibit endotoxin-induced TNF-alpha production in humans. FASEB J. 2003 May;17(8):884-6. doi: 10.1096/fj.02-0670fje. Epub 2003 Mar 5. PMID 12626436
- [Background] Steensberg A, Fischer CP, Keller C, Moller K, Pedersen BK. IL-6 enhances plasma IL-1ra, IL-10, and cortisol in humans. Am J Physiol Endocrinol Metab. 2003 Aug;285(2):E433-7. doi: 10.1152/ajpendo.00074.2003. PMID 12857678
- [Background] Tisdale MJ. Mechanisms of cancer cachexia. Physiol Rev. 2009 Apr;89(2):381-410. doi: 10.1152/physrev.00016.2008. PMID 19342610
- [Background] von Haehling S, Anker SD. Cachexia as a major underestimated and unmet medical need: facts and numbers. J Cachexia Sarcopenia Muscle. 2010 Sep;1(1):1-5. doi: 10.1007/s13539-010-0002-6. Epub 2010 Oct 26. PMID 21475699
- [Background] Zammit PS, Partridge TA, Yablonka-Reuveni Z. The skeletal muscle satellite cell: the stem cell that came in from the cold. J Histochem Cytochem. 2006 Nov;54(11):1177-91. doi: 10.1369/jhc.6R6995.2006. Epub 2006 Aug 9. PMID 16899758
- [Background] Zoico E, Roubenoff R. The role of cytokines in regulating protein metabolism and muscle function. Nutr Rev. 2002 Feb;60(2):39-51. doi: 10.1301/00296640260085949. PMID 11852969
- [Background] Trost SG, Owen N, Bauman AE, Sallis JF, Brown W. Correlates of adults' participation in physical activity: review and update. Med Sci Sports Exerc. 2002 Dec;34(12):1996-2001. doi: 10.1097/00005768-200212000-00020. PMID 12471307
- [Background] Gibala MJ, Gillen JB, Percival ME. Physiological and health-related adaptations to low-volume interval training: influences of nutrition and sex. Sports Med. 2014 Nov;44 Suppl 2(Suppl 2):S127-37. doi: 10.1007/s40279-014-0259-6. PMID 25355187
- [Background] Gillen JB, Gibala MJ. Is high-intensity interval training a time-efficient exercise strategy to improve health and fitness? Appl Physiol Nutr Metab. 2014 Mar;39(3):409-12. doi: 10.1139/apnm-2013-0187. Epub 2013 Sep 27. PMID 24552392
- [Background] Gillen JB, Percival ME, Ludzki A, Tarnopolsky MA, Gibala MJ. Interval training in the fed or fasted state improves body composition and muscle oxidative capacity in overweight women. Obesity (Silver Spring). 2013 Nov;21(11):2249-55. doi: 10.1002/oby.20379. Epub 2013 May 31. PMID 23723099
- [Background] Allison MK, Baglole JH, Martin BJ, Macinnis MJ, Gurd BJ, Gibala MJ. Brief Intense Stair Climbing Improves Cardiorespiratory Fitness. Med Sci Sports Exerc. 2017 Feb;49(2):298-307. doi: 10.1249/MSS.0000000000001188. PMID 28009784
- [Background] Gist NH, Freese EC, Cureton KJ. Comparison of responses to two high-intensity intermittent exercise protocols. J Strength Cond Res. 2014 Nov;28(11):3033-40. doi: 10.1519/JSC.0000000000000522. PMID 24832968
- [Background] Sperlich B, Wallmann-Sperlich B, Zinner C, Von Stauffenberg V, Losert H, Holmberg HC. Functional High-Intensity Circuit Training Improves Body Composition, Peak Oxygen Uptake, Strength, and Alters Certain Dimensions of Quality of Life in Overweight Women. Front Physiol. 2017 Apr 3;8:172. doi: 10.3389/fphys.2017.00172. eCollection 2017. PMID 28420999
- [Background] Emberts T, Porcari J, Dobers-Tein S, Steffen J, Foster C. Exercise intensity and energy expenditure of a tabata workout. J Sports Sci Med. 2013 Sep 1;12(3):612-3. eCollection 2013. No abstract available. PMID 24137082
- [Derived] Limirio LS, Rossato LT, Barbosa CD, Teixeira KRC, Nahas PC, de Branco FMS, Martins FM, Nomelini RS, Murta EFC, Orsatti FL, de Oliveira EP. Body Mass Index, waist circumference or sagittal abdominal diameter: Which parameter is better correlated with body fat changes in postmenopausal women after combined training protocol? Clin Nutr ESPEN. 2020 Aug;38:192-195. doi: 10.1016/j.clnesp.2020.05.004. Epub 2020 May 30. PMID 32690157
- [Derived] Nunes PRP, Martins FM, Souza AP, Carneiro MAS, Nomelini RS, Michelin MA, Murta EFC, de Oliveira EP, Orsatti FL. Comparative effects of high-intensity interval training with combined training on physical function markers in obese postmenopausal women: a randomized controlled trial. Menopause. 2019 Nov;26(11):1242-1249. doi: 10.1097/GME.0000000000001399. PMID 31479035
- [Derived] Martins FM, de Paula Souza A, Nunes PRP, Michelin MA, Murta EFC, Resende EAMR, de Oliveira EP, Orsatti FL. High-intensity body weight training is comparable to combined training in changes in muscle mass, physical performance, inflammatory markers and metabolic health in postmenopausal women at high risk for type 2 diabetes mellitus: A randomized controlled clinical trial. Exp Gerontol. 2018 Jul 1;107:108-115. doi: 10.1016/j.exger.2018.02.016. Epub 2018 Feb 19. PMID 29471132